CLINICAL TRIAL: NCT02485574
Title: Prospective, Observational Study of Anterior Bridging Cage Augmented With Bone Substitute Versus Localized Autobone in Transforaminal Lumbar Interbody Arthrodesis
Brief Title: Anterior Bridging Cage With Bone Substitute Versus Localized Autobone in Transforaminal Lumbar Interbody Arthrodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zenoss Co, Ltd (Other)
Responsible Party: Principal Investigator, Kwang Sup Song, Professor, Zenoss Co, Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSong
Record Dates: First submitted 2015-06-12; First posted 2015-06-30 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Stenosis; Fusion of Spine (Disease)
Keywords: Bone bridging; Arthrodesis; Lumbar; Cage
MeSH Terms: conditions — Constriction, Pathologic; Disease; Ankylosis | interventions — Durapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left cage- auto bone (Experimental): At the operated segment, left cage was filled with auto bone only. We evaluated bone bridging between inside and outside the cage in transforaminal lumbar interbody arthrodesis.
  Interventions: Procedure: transforaminal lumbar interbody arthrodesis
- Right cage- auto local bone mixed with β-calcium phosphate + hydroxyapatite (Experimental): At the operated segment, right cage was filled with auto local bone mixed with β-calcium phosphate + hydroxyapatite. We evaluated bone bridging between inside and outside the cage in transforaminal lumbar interbody arthrodesis.
  Interventions: Procedure: transforaminal lumbar interbody arthrodesis

INTERVENTIONS:
Procedure: transforaminal lumbar interbody arthrodesis — Anterior bridging cages augmented with auto bone plus β-calcium phosphate + hydroxyapatite in right side of disc space and anterior bridging cages augmented with auto bone in left side of disc space in transforaminal lumbar interbody arthrodesis.
  Other Names: β-calcium phosphate + hydroxyapatite (OSTEON 2, Genoss); Auto-local bone

SUMMARY:
The purpose of this study is to evaluation for the pattern of bone bridging of patients who undergo transforaminal lumbar interbody arthrodesis, the investigators hypothesize that auto local bone mixed with β-calcium phosphate + hydroxyapatite (OSTEON 2, Genoss) is not inferior to auto local bone only. In addition, the investigators will analyze anterior new bone bridging pattern between anterior bridging cage newly developed and grafted bone in anterior disc space.

DETAILED DESCRIPTION:
A single center, observational, single arm study to evaluate the efficacy of auto local bone mixed with β-calcium phosphate + hydroxyapatite using interbody fusion assessment on multi-axial CT scan. Its active comparator is auto local bone.

Anterior bridging bone between anterior grafted bone and inserted cage will be assessed by using newly developed anterior bridging cage as well as interbody bone bridging between two vertebral bodies on multi-axial reconstructed CT scan.

The patients undergoes arthrodesis surgery will have two cages, one augmented with auto local bone will be located at left side of disc space and the other cage augmented with auto local bone mixed with β-calcium phosphate + hydroxyapatite at right side of disc space.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need lumbar interbody fusion in Degenerative spine disease on L1-S1(Spinal stenosis, HIVD and internal derangement of disk, spine instability)
* Patients who have no communication problems
* Patients who are willing to visit the hospital for any follow-up assessment
* Patients who voluntarily sign on a written consent

Exclusion Criteria:

* Patients who have infection
* Patients who have bleeding disorders
* Patients who have immunosuppressed disease
* Patients who can't sign on consent form
* Patients who are in pregnancy or breast feeding
* Patients who have severe osteoporosis
* Patients who can't take general surgery because of severe liver disease or decreased renal function
* Patients who have acute spinal injury, spinal tumor or inflammatory spinal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Sup Song, M.D., PhD, Principal Investigator — Chung-Ang University
Locations (1):
- Kwang Sup Song, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy DR, Hurwitz EL, Gregory A, Clary R. A nonsurgical approach to the management of patients with cervical radiculopathy: a prospective observational cohort study. J Manipulative Physiol Ther. 2006 May;29(4):279-87. doi: 10.1016/j.jmpt.2006.03.005. PMID 16690382
- [Background] SMITH GW, ROBINSON RA. The treatment of certain cervical-spine disorders by anterior removal of the intervertebral disc and interbody fusion. J Bone Joint Surg Am. 1958 Jun;40-A(3):607-24. No abstract available. PMID 13539086
- [Background] CLOWARD RB. The anterior approach for removal of ruptured cervical disks. J Neurosurg. 1958 Nov;15(6):602-17. doi: 10.3171/jns.1958.15.6.0602. No abstract available. PMID 13599052
- [Background] Coric D, Branch CL Jr, Jenkins JD. Revision of anterior cervical pseudoarthrosis with anterior allograft fusion and plating. J Neurosurg. 1997 Jun;86(6):969-74. doi: 10.3171/jns.1997.86.6.0969. PMID 9171175
- [Background] Savolainen S, Rinne J, Hernesniemi J. A prospective randomized study of anterior single-level cervical disc operations with long-term follow-up: surgical fusion is unnecessary. Neurosurgery. 1998 Jul;43(1):51-5. doi: 10.1097/00006123-199807000-00032. PMID 9657188
- [Background] Shapiro S. Banked fibula and the locking anterior cervical plate in anterior cervical fusions following cervical discectomy. J Neurosurg. 1996 Feb;84(2):161-5. doi: 10.3171/jns.1996.84.2.0161. PMID 8592216
- [Background] Wang JC, McDonough PW, Endow KK, Delamarter RB. Increased fusion rates with cervical plating for two-level anterior cervical discectomy and fusion. Spine (Phila Pa 1976). 2000 Jan;25(1):41-5. doi: 10.1097/00007632-200001010-00009. PMID 10647159
- [Background] Zoega B, Karrholm J, Lind B. Plate fixation adds stability to two-level anterior fusion in the cervical spine: a randomized study using radiostereometry. Eur Spine J. 1998;7(4):302-7. doi: 10.1007/s005860050079. PMID 9765038
- [Background] Abd-Alrahman N, Dokmak AS, Abou-Madawi A. Anterior cervical discectomy (ACD) versus anterior cervical fusion (ACF), clinical and radiological outcome study. Acta Neurochir (Wien). 1999;141(10):1089-92. doi: 10.1007/s007010050487. PMID 10550654
- [Background] An HS, Simpson JM, Glover JM, Stephany J. Comparison between allograft plus demineralized bone matrix versus autograft in anterior cervical fusion. A prospective multicenter study. Spine (Phila Pa 1976). 1995 Oct 15;20(20):2211-6. PMID 8545714
- [Background] Bishop RC, Moore KA, Hadley MN. Anterior cervical interbody fusion using autogeneic and allogeneic bone graft substrate: a prospective comparative analysis. J Neurosurg. 1996 Aug;85(2):206-10. doi: 10.3171/jns.1996.85.2.0206. PMID 8755747
- [Background] Cauthen JC, Kinard RE, Vogler JB, Jackson DE, DePaz OB, Hunter OL, Wasserburger LB, Williams VM. Outcome analysis of noninstrumented anterior cervical discectomy and interbody fusion in 348 patients. Spine (Phila Pa 1976). 1998 Jan 15;23(2):188-92. doi: 10.1097/00007632-199801150-00008. PMID 9474724
- [Background] Geisler FH, Caspar W, Pitzen T, Johnson TA. Reoperation in patients after anterior cervical plate stabilization in degenerative disease. Spine (Phila Pa 1976). 1998 Apr 15;23(8):911-20. doi: 10.1097/00007632-199804150-00013. PMID 9580959
- [Background] Hacker RJ, Cauthen JC, Gilbert TJ, Griffith SL. A prospective randomized multicenter clinical evaluation of an anterior cervical fusion cage. Spine (Phila Pa 1976). 2000 Oct 15;25(20):2646-54; discussion 2655. doi: 10.1097/00007632-200010150-00017. PMID 11034651
- [Background] Lofgren H, Johannsson V, Olsson T, Ryd L, Levander B. Rigid fusion after cloward operation for cervical disc disease using autograft, allograft, or xenograft: a randomized study with radiostereometric and clinical follow-up assessment. Spine (Phila Pa 1976). 2000 Aug 1;25(15):1908-16. doi: 10.1097/00007632-200008010-00008. PMID 10908933
- [Background] Lowery GL, McDonough RF. The significance of hardware failure in anterior cervical plate fixation. Patients with 2- to 7-year follow-up. Spine (Phila Pa 1976). 1998 Jan 15;23(2):181-6; discussion 186-7. doi: 10.1097/00007632-199801150-00006. PMID 9474723
- [Background] Tribus CB, Corteen DP, Zdeblick TA. The efficacy of anterior cervical plating in the management of symptomatic pseudoarthrosis of the cervical spine. Spine (Phila Pa 1976). 1999 May 1;24(9):860-4. doi: 10.1097/00007632-199905010-00005. PMID 10327506
- [Background] Gercek E, Arlet V, Delisle J, Marchesi D. Subsidence of stand-alone cervical cages in anterior interbody fusion: warning. Eur Spine J. 2003 Oct;12(5):513-6. doi: 10.1007/s00586-003-0539-6. Epub 2003 Jun 21. PMID 12827473
- [Background] Bagby GW. Arthrodesis by the distraction-compression method using a stainless steel implant. Orthopedics. 1988 Jun;11(6):931-4. doi: 10.3928/0147-7447-19880601-13. PMID 3387340
- [Background] DeBowes RM, Grant BD, Bagby GW, Gallina AM, Sande RD, Ratzlaff MH. Cervical vertebral interbody fusion in the horse: a comparative study of bovine xenografts and autografts supported by stainless steel baskets. Am J Vet Res. 1984 Jan;45(1):191-9. PMID 6367560
- [Background] Wilke HJ, Kettler A, Goetz C, Claes L. Subsidence resulting from simulated postoperative neck movements: an in vitro investigation with a new cervical fusion cage. Spine (Phila Pa 1976). 2000 Nov 1;25(21):2762-70. doi: 10.1097/00007632-200011010-00008. PMID 11064521
- [Background] Toth JM, Wang M, Estes BT, Scifert JL, Seim HB 3rd, Turner AS. Polyetheretherketone as a biomaterial for spinal applications. Biomaterials. 2006 Jan;27(3):324-34. doi: 10.1016/j.biomaterials.2005.07.011. Epub 2005 Aug 22. PMID 16115677
- [Background] Kurtz SM, Devine JN. PEEK biomaterials in trauma, orthopedic, and spinal implants. Biomaterials. 2007 Nov;28(32):4845-69. doi: 10.1016/j.biomaterials.2007.07.013. Epub 2007 Aug 7. PMID 17686513
- [Background] Yao C, Storey D, Webster TJ. Nanostructured metal coatings on polymers increase osteoblast attachment. Int J Nanomedicine. 2007;2(3):487-92. PMID 18019846
- [Background] Han CM, Lee EJ, Kim HE, Koh YH, Kim KN, Ha Y, Kuh SU. The electron beam deposition of titanium on polyetheretherketone (PEEK) and the resulting enhanced biological properties. Biomaterials. 2010 May;31(13):3465-70. doi: 10.1016/j.biomaterials.2009.12.030. Epub 2010 Feb 13. PMID 20153890
- [Background] Cho DY, Lee WY, Sheu PC, Chen CC. Cage containing a biphasic calcium phosphate ceramic (Triosite) for the treatment of cervical spondylosis. Surg Neurol. 2005 Jun;63(6):497-503; discussion 503-4. doi: 10.1016/j.surneu.2004.10.016. PMID 15936361
- [Background] Kast E, Derakhshani S, Bothmann M, Oberle J. Subsidence after anterior cervical inter-body fusion. A randomized prospective clinical trial. Neurosurg Rev. 2009 Apr;32(2):207-14; discussion 214. doi: 10.1007/s10143-008-0168-y. Epub 2008 Sep 17. PMID 18797946
- [Background] Kulkarni AG, Hee HT, Wong HK. Solis cage (PEEK) for anterior cervical fusion: preliminary radiological results with emphasis on fusion and subsidence. Spine J. 2007 Mar-Apr;7(2):205-9. doi: 10.1016/j.spinee.2006.03.002. Epub 2006 Nov 17. PMID 17321970
- [Background] Cho DY, Liau WR, Lee WY, Liu JT, Chiu CL, Sheu PC. Preliminary experience using a polyetheretherketone (PEEK) cage in the treatment of cervical disc disease. Neurosurgery. 2002 Dec;51(6):1343-49; discussion 1349-50. PMID 12445338
- [Background] Kandziora F, Pflugmacher R, Scholz M, Schnake K, Putzier M, Khodadadyan-Klostermann C, Haas NP. Treatment of traumatic cervical spine instability with interbody fusion cages: a prospective controlled study with a 2-year follow-up. Injury. 2005 Jul;36 Suppl 2:B27-35. doi: 10.1016/j.injury.2005.06.012. PMID 15993115

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants - Single Group: Consecutive patients with spinal stenosis or spondylolisthesis who planned to undergo single-level transforaminal lumbar interbody fusion (TLIF) with pedicle screw fixation were included. After disc preparation following bilateral decompression with facetectomies, extra-cage bone grafting, consisting of half- mixed each 6 cc of local autobone and synthetic bone, was performed on the prepared anterior disc space bilaterally; then, bilateral cages with different graft compositions (left cage: filled with local autobone, right cage: filled with local autobone þ synthetic bone) were inserted in "same segment". We compared the anterior bone bridging patterns of two cages "at single operated segment" in each patient.
Period: Overall Study
Arm/Group | All Study Participants - Single Group
Started | 69
Completed | 65
Not Completed | 4
Not completed — dropped out because they failed to undergo CT scan at postoperative 12 months | 4

BASELINE CHARACTERISTICS:
Population: 69 patients were enrolled. Out of the total study participants, 4 patients dropped out because they failed to undergo CT scan at postoperative 12 months.
Groups:
- All Study Participants: Consecutive patients with spinal stenosis or spondylolisthesis who planned to undergo single-level transforaminal lumbar interbody fusion (TLIF) with pedicle screw fixation were included. After disc preparation following bilateral decompression with facetectomies, extra-cage bone grafting, consisting of half- mixed each 6 cc of local autobone and synthetic bone, was performed on the prepared anterior disc space bilaterally; then, bilateral cages with different graft compositions (left cage: filled with local autobone, right cage: filled with local autobone þ synthetic bone) were inserted. We compared the anterior bone bridging patterns of two cages in each patient.
Arm/Group | All Study Participants
Number analyzed (Participants) | 69
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66.7 [65.7 to 67.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 65
body mass index [Mean (Inter-Quartile Range); unit: kg/m^2] | 25.3 [24.3 to 26.3]

OUTCOME MEASURES:

1. Primary Outcome: InCBB of Both Cages
Description: We used the concept of InCBB (intra-cage bridging bone) to evaluate the fusion status. InCBB was defined as the bridging bone between the upper and lower vertebrae through the void of the cage(s) and divided into right (Rt.) and left (Lt.) InCBB according to the cage position. We graded bridging scores from 0 to 2 based on the degree of completion of the bridging bone in InCBBs (grade 0: no bridging at the superior and inferior endplates; grade 1: incomplete bridging; bridging at the superior or inferior endplate, but with a clear radiolucent line; grade 2: complete bridging).
Time Frame: 12 month postoperatively
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Left Cage- Auto Bone: Consecutive patients with spinal stenosis or spondylolisthesis who planned to undergo single-level transforaminal lumbar interbody fusion (TLIF) with pedicle screw fixation were included. After disc preparation following bilateral decompression with facetectomies, extra-cage bone grafting, consisting of half- mixed each 6 cc of local autobone and synthetic bone, was performed on the prepared anterior disc space bilaterally. At the operated segment, left cage was filled with auto bone only.
- Right Cage- Auto Local Bone Mixed With β-calcium Phosphate + Hydroxyapatite: Consecutive patients with spinal stenosis or spondylolisthesis who planned to undergo single-level transforaminal lumbar interbody fusion (TLIF) with pedicle screw fixation were included. After disc preparation following bilateral decompression with facetectomies, extra-cage bone grafting, consisting of half- mixed each 6 cc of local autobone and synthetic bone, was performed on the prepared anterior disc space bilaterally. At the operated segment, right cage was filled with auto local bone mixed with β-calcium phosphate + hydroxyapatite.
Arm/Group | Left Cage- Auto Bone | Right Cage- Auto Local Bone Mixed With β-calcium Phosphate + Hydroxyapatite
Number analyzed (Participants) | 65 | 65
score on a scale | 1.48 [1.44 to 1.53] | 1.43 [1.39 to 1.48]

2. Secondary Outcome: ABB (Anterior Bone Bridging) Between Cage and Anterior Grafted Bone
Description: We defined ABB as the bridging bone between the extra-cage grafted bone and intra-cage grafted bone through the holes in each cage. Since the cages used in this study each have 4 anterior holes, there can be a minimum of 0 and a maximum of 8 ABBs in a patient.
Time Frame: 12 month postoperatively
Measure: Mean (95% Confidence Interval); unit: number of anterior holes
Groups:
- Left Cage- Auto Bonegroup: Consecutive patients with spinal stenosis or spondylolisthesis who planned to undergo single-level transforaminal lumbar interbody fusion (TLIF) with pedicle screw fixation were included. After disc preparation following bilateral decompression with facetectomies, extra-cage bone grafting, consisting of half- mixed each 6 cc of local autobone and synthetic bone, was performed on the prepared anterior disc space bilaterally. At the operated segment, left cage was filled with auto bone only.
Arm/Group | Left Cage- Auto Bonegroup | Right Cage- Auto Local Bone Mixed With β-calcium Phosphate + Hydroxyapatite
Number analyzed (Participants) | 65 | 65
number of anterior holes | 1.80 [1.68 to 1.92] | 1.85 [1.72 to 1.97]

3. Other Pre Specified Outcome: ODI Change (Preoperative ODI Score - Postoperative 1 Year ODI Score)
Description: The Oswestry Disability Index (ODI) is an index used by clinicians and researchers to quantify disability for low back pain.
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: postoperative 1 year
Population: Of the total 65 patients, 56 were classified as having interbody fusion, and 9 were classified as not having interbody fusion.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Interbody Fused Group: We determined the interbody fusion as "in cases with at least one or more complete InCBB and/or ExCBB on both sagittal and coronal views simultaneously without subsidence".
  This group was classified as having achieved interbody fusion.
- Interbody Unfused Group: We determined the interbody fusion in cases with at least one or more complete InCBB and/or ExCBB on both sagittal and coronal views simultaneously without subsidence.
  This group was classified as not having achieved interbody fusion.
Arm/Group | Interbody Fused Group | Interbody Unfused Group
Number analyzed (Participants) | 56 | 9
score on a scale | 45.53 [43.29 to 47.90] | 35.19 [32.92 to 37.40]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Left Cage- Auto Bone | Right Cage- Auto Local Bone Mixed With β-calcium Phosphate + Hydroxyapatite
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

LIMITATIONS AND CAVEATS:
Suggested criterios can only be used for interbody fusion evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT02485574/Prot_SAP_000.pdf